CLINICAL TRIAL: NCT02798939
Title: Evaluation of Lactoferrin, Procalcitonin and Aution® Urine Dipsticks for the Diagnosis of Spontaneous Bacterial Peritonitis in Cirrhotic Patients
Status: Terminated | Type: Observational
Why Stopped: investigator choice
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: AOL09-NGUYEN-KHAC
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Liver Cirrhosis
Keywords: spontaneous bacterial peritonitis; lactoferrin; procalcitonin; Aution® urine dipsticks
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — ascitic fluid

GROUPS / COHORTS (1):
- cirrhotic patients

SUMMARY:
Bacterial infections are a major cause of mortality in cirrhotic patients in the context of gastrointestinal bleeding or spontaneous bacterial peritonitis (SBP). Rapid diagnosis of SBP is therefore an important research goal because the gold standard neutrophil count in ascitic fluid cannot be performed 24 hours a day in all healthcare structures. The use of urine dipsticks in ascites cannot be recommended at the present time due to their insufficient sensitivity with an unacceptable risk of false-negatives in the context of a fatal disease for which effective antibiotic therapy is available. Ascitic fluid lactoferrin assay has recently been demonstrated to be a very good diagnostic test for SBP. The investigators plan to conduct a prospective study on lactoferrin as well as procalcitonin (PCT) to determine the best laboratory test(s) for the rapid, automated diagnosis of SBP. These tests will be compared with the Aution® urine dipstick, which has been shown to present better diagnostic sensitivity than the Multistix® dipstick . This single-centre study (Amiens University Hospital) will be performed in the context of routine clinical practice on ascitic fluid that is usually incinerated.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years, not unable major
* Cirrhosis diagnosed by liver histology (or a non-invasive test , biological, or Fibrotest Fibrometer , or physical Fibroscan® ) , or a set of clinical, laboratory , ultrasound and endoscopy .
* Presence of ascites puncture in the clinical part of routine care

Exclusion Criteria:

* Ascites noncirrhotic origins : heart , nephrotic syndrome, peritoneal dialysis, tuberculosis, cancer peritoneal carcinomatosis , acute and chronic pancreatitis
* surgical peritonitis by perforation of hollow organ
* Haemoperitoneum pure or associated with ascites.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhotic patients requiring ascitic fluid aspiration, routine clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2010-03-01 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2017-02-14 (Actual)

PRIMARY OUTCOMES:
diagnostic performances of lactoferrin | D0
diagnostic performances of PCT | D0
diagnostic performances of Aution® urine dipstick | D0

CONTACTS AND LOCATIONS:
Overall Officials: Eric NGUYEN KHAC, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France